CLINICAL TRIAL: NCT02819622
Title: Persona of Central Serous Chorioretinopathy
Acronym: CSCR
Status: Completed | Type: Observational
Sponsor: Rafic Hariri University Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Mansour, MD, Clinical Professor, AUB, Chair, Department of Opthalmology, Rafic Hariri Hospital, Rafic Hariri University Hospital
Other Study IDs: INV-2014-204
Record Dates: First submitted 2016-06-14; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Personality Type

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: control (no disease)
- central serous retinopathy group: Central serous retinopathy (with CSCR disease) by exam and OCT

SUMMARY:
Purpose: Central serous retinopathy (CSCR) is characterized by macular detachment due to thickened choroid mostly affecting young men under perceived stress. While most previous studies in CSCR have been retrospective and have focused on a single facet of the patient's personality, the investigators conducted a prospective intercontinental controlled study to analyze the multifaceted personality profile in CSCR.

Design: Prospective interview. Participants and Controls: Subjects with CSCR consented to participate in a questionnaire. Controls not having retinal disease were recruited from the same clinic.

Main Outcome Measures: The main parameters registered were presence of stress, daily number of cups caffeine intake, personality traits (Type A; obsessive-compulsive; aggressive).

Methods: The interview consisted of a 60-item questionnaire. Recruitment of participants was from January 2015 to February 2016. Controls were matched for age, gender and race. Statistical analyses were done using univariate and multivariate analysis.

DETAILED DESCRIPTION:
Central serous chorioretinopathy (CSCR) characterized by serous macular detachment is the fourth most common retinal disease after age-related macular degeneration, diabetic retinopathy and retinal vein occlusion. In a population-based retrospective cohort and case control study in Olmsted county, Minnesota, USA, Kitzmann et al4 reported a mean age-adjusted incidence of 9.9 (95% confidence interval [CI] 7.4-12.4) per 100, 000 in men, and 1.7 (95% CI 0.7-2.7) in women. The mean age of onset of CSCR appears between 41 and 45 years5. The disease affects various racial groups5-8 and occasionally can be familial9. The pathogenesis remains poorly understood and currently the exudation is thought to result from hyper-permeable choroid secondary to venous stasis, ischemia, or inflammation2. Because of lack of proper animal models and lack of definite cure, clinical research has focused on risk factors such as stress, corticosteroid intake, and type A personality. Different hospital-based studies yielded different risk factors. Epidemiologic studies failed to ascertain many of these risk factors. Due to different methodology (retrospective vs. prospective case-control studies; selection of controls; questionnaire vs. interview by physician assistant vs. interview by physician) and focus on single risk factors in the literature, the investigators designed a study that targets a vast number of known or potential risk factors in various collaborative centers and compare it to results reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

* clinical evidence by fluorescein angiography and OCT of CSCR disease
* willingness to undergo long interview
* ability to sign an informed consent

Exclusion Criteria:

* severe systemic hypertension
* eclampsia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with central serous retinopathy
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
personality type | through study completion, an average of 1 year
  one interview by the ophthalmologist himself

CONTACTS AND LOCATIONS:
Overall Officials: ahmad mansour, md, Principal Investigator — RHUH
Locations (1):
- Rafic Hariri University Hospital, Beirut, South Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
publication and excel sheet

REFERENCES:
- [Background] Liu B, Deng T, Zhang J. RISK FACTORS FOR CENTRAL SEROUS CHORIORETINOPATHY: A Systematic Review and Meta-Analysis. Retina. 2016 Jan;36(1):9-19. doi: 10.1097/IAE.0000000000000837. PMID 26710181
- [Background] Daruich A, Matet A, Dirani A, Bousquet E, Zhao M, Farman N, Jaisser F, Behar-Cohen F. Central serous chorioretinopathy: Recent findings and new physiopathology hypothesis. Prog Retin Eye Res. 2015 Sep;48:82-118. doi: 10.1016/j.preteyeres.2015.05.003. Epub 2015 May 27. PMID 26026923
- [Background] Sacca SC, Vagge A, Pulliero A, Izzotti A. Helicobacter pylori infection and eye diseases: a systematic review. Medicine (Baltimore). 2014 Dec;93(28):e216. doi: 10.1097/MD.0000000000000216. PMID 25526440
- [Background] Mateo-Montoya A, Mauget-Fayse M. Helicobacter pylori as a risk factor for central serous chorioretinopathy: Literature review. World J Gastrointest Pathophysiol. 2014 Aug 15;5(3):355-8. doi: 10.4291/wjgp.v5.i3.355. PMID 25133035